CLINICAL TRIAL: NCT07113977
Title: Clinical Study of a Novel Humanized CD70-Targeted CAR-T Cell Incorporating TLR2 for Advanced Renal Cell Carcinoma Therapy
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Wei Guan (Other)
Responsible Party: Sponsor-Investigator, Wei Guan, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJ-IRB202502144
Record Dates: First submitted 2025-07-24; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Advanced Renal Cell Carcinoma
Keywords: CD70; CAR-T; Advanced renal cell carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental)
  Interventions: Biological: CAR-T(CD70)

INTERVENTIONS:
Biological: CAR-T(CD70) — In this clinical study, participants with advanced renal cell carcinoma will receive a novel humanized CD70-targeted CAR-T-cell product that incorporates the TLR2 co-stimulatory domain. Peripheral blood mononuclear cells will be collected from each subject, genetically modified to express the CAR construct, and expanded ex vivo; after passing multiple quality-control assays, the CAR-T cells will be administered intratumorally under CT guidance at the pre-specified dose. Following treatment, the efficacy and safety of CD70-directed CAR-T-cell therapy will be comprehensively assessed through clinical symptom evaluations, quality-of-life questionnaires, biomarker analyses, laboratory tests, imaging studies, adverse-event monitoring, and long-term follow-up.

SUMMARY:
In this clinical study, participants with advanced renal cell carcinoma will receive a novel humanized CD70-targeted CAR-T-cell product that incorporates the TLR2 co-stimulatory domain. Peripheral blood mononuclear cells will be collected from each subject, genetically modified to express the CAR construct, and expanded ex vivo; after passing multiple quality-control assays, the CAR-T cells will be infused at the pre-specified dose. Post-infusion, the efficacy and safety of CD70-directed CAR-T-cell therapy will be systematically evaluated using clinical symptom assessments, quality-of-life questionnaires, biomarker analyses, laboratory tests, imaging studies, adverse-event monitoring, and long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 1. Voluntary participation with written informed consent provided by the patient or legally authorized representative;
* 2.Age 18-75 years (inclusive) at the time of consent, regardless of sex;
* 3.Advanced-stage renal cell carcinoma (RCC) with no curative treatment options, who have received ≥1 prior line of therapy and meet one or more of the following:

  1. Recurrence after first-line or later-line treatment(s).
  2. Progression or persistent progression following prior therapy;
* 4.Histopathologically confirmed advanced RCC per WHO 2016 classification, with at least one measurable lesion evaluable by CT or MRI;
* 5.CD70 positivity in tumor tissue confirmed by immunohistochemistry (IHC);
* 6.Adequate organ function: Hepatic: ALT/AST <3× ULN and total bilirubin ≤34.2 μmol/L. Renal: Creatinine clearance (Cockcroft-Gault) ≥60 mL/min. Pulmonary: Oxygen saturation ≥95% with no active pulmonary infection. Cardiac: LVEF ≥50%, no significant pericardial effusion, and no clinically relevant ECG abnormalities;
* 7.Contraception: Women of childbearing potential must have a negative pregnancy test (urine/serum) at screening and agree to use effective contraception for ≥1 year post-infusion.

Men with partners of childbearing potential must use barrier contraception for ≥1 year post-infusion;

* 8.Performance status: ECOG score 0-3;
* 9.Life expectancy >3 months;
* 10.Willingness to comply with leukapheresis, medical assessments, and follow-up visits.

Exclusion Criteria:

* 1.Pregnant or lactating women;
* 2.Uncontrolled fungal, bacterial, Treponema pallidum, viral, or other infections;
* 3.Active hepatitis: HBV DNA >500 IU/mL. Positive HCV RNA (confirmed by repeat testing);
* 4.HIV infection, known acquired immunodeficiency syndrome (AIDS), or syphilis infection;
* 5.Prior gene therapy of any form;
* 6.History of severe allergic reactions to biologics (including antibiotics), antibodies, cytokines, or other macromolecular agents;
* 7.Clinically significant CNS disorders: epilepsy, paresis, aphasia, stroke, severe traumatic brain injury, dementia, Parkinson's disease, cerebellar disorders, organic brain syndrome;
* 8.Uncontrolled psychiatric illness;
* 9.Substance abuse/addiction;
* 10.Prohibited medications/treatments: Corticosteroids: ≥2 mg/kg prednisone (or equivalent >20 mg/day) within 2 weeks before leukapheresis.

Chemo/radiotherapy: Anti-tumor radiotherapy or salvage chemotherapy within 3 weeks before leukapheresis.

Immunosuppressants: Use within 4 weeks before leukapheresis. Other trials/major surgery: Participation in another clinical trial or major non-diagnostic surgery within 4 weeks before leukapheresis.

Specific agents: Alemtuzumab within 6 months, or clofarabine/cladribine within 3 months before leukapheresis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Immune Effector Cell-Associated Neurotoxicity Syndrome（ICANS） | in 6 months
  To assess the number and severity of ICANS after treatment according to the ASTCT criteria
Cytokine Release Syndrome（CRS） | in 6 months
  To assess the number and severity of CRS after treatment according to the ASTCT criteria
Objective response rate (ORR) | 1 month, 6 months, and 1 year
  Objective response rate (ORR) will be assessed by imaging at 1 month, 6 months, and 1 year post-CAR-T infusion.

SECONDARY OUTCOMES:
Progression-Free Survival（PFS） | The time from the start of treatment to disease progression, up to a maximum of 36 months.
Overall Survival（OS） | The time from the start of treatment to death, up to a maximum of 36 months.
Adverse Events | in six months
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

IPD SHARING:
Plan to Share IPD: No